CLINICAL TRIAL: NCT00388674
Title: Randomized, Observational Study of Entecavir to Assess Long-term Outcomes Associated With Nucleoside/Nucleotide Monotherapy for Patients With Chronic HBV Infection: The REALM Study
Brief Title: Study of Entecavir in Patients With Chronic Hepatitis B Virus (HBV) Infection
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI463-080
Record Dates: First submitted 2006-10-04; First posted 2006-10-17 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-10

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B Virus
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — buccal
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A
  Interventions: Drug: entecavir
- B
  Interventions: Drug: Other anti-HBV medication

INTERVENTIONS:
Drug: entecavir — Tablets / Oral Solution, Oral, ETV = 0.5 mg - 1 mg, once daily, Investigator/Patient decision
  Other Names: Baraclude; BMS-200475
  Groups: A
Drug: Other anti-HBV medication — Tablets / Oral Solution, Oral, depends on chosen active comparator, depends on chosen active comparator, Investigator/Patient decision
  Groups: B

SUMMARY:
The purpose of this study is to prospectively assess the long-term outcomes (benefits and risks) associated with entecavir (ETV) therapy as compared to other antivirals approved for the treatment of chronic HBV infection. For the China substudy, patients randomized to entecavir will have safety and efficacy assessments performed during the first year of the study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HBV infection
* HBV nucleoside/tide-naive or -experienced
* Patients who, in opinion of investigator, are appropriate for initiating or modifying their HBV therapy and who are appropriate for a treatment regimen comprised of nucleoside/tide monotherapy with either ETV or another standard of care HBV nucleoside/tide analogue
* Age 16 and older or minimum age required in a given country

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Patients who, in the opinion of the investigator, are expected to have a liver transplant-free survival of less than one year
* Patients who, in the opinion of the investigator, are virologically controlled on their current treatment regimen and clinically responding to treatment, unless the regimen needs to be modified for medication intolerance
* Coinfection with HIV
* History of malignant neoplasm(s), including hepatocellular carcinoma (HCC) and carcinoma in situ (CIS), but excluding non-melanoma skin cancers
* Patients with chronic renal insufficiency, defined as a creatinine clearance < 50 ml/min who do not have either of the following means of dose reducing ETV:

  i. an approved country-specific ETV label which includes the extended interval ETV dose modification method and/or ii. an approved country specific label for the ETV oral solution AND access to the oral solution
* History of dysplastic liver nodules
* Known history of allergy to nucleoside/tide analogues
* Prior or current treatment with entecavir
* An investigator proposed study regimen which will include only interferon-alfa
* An investigator proposed study regimen of combination (two or more) HBV nucleoside/tide analogues

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic hepatitis B patients receiving nucleoside therapy
Sampling Method: Non-Probability Sample
Enrollment: 12522 (Actual)
Dates: Start 2006-12-18 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2016-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Chair — Bristol-Myers Squibb
Locations (220):
- United States (20):
  - Scti Research Foundation, Coronado, California
  - Cedars-Sinai Comprehensive Transplant Center, Los Angeles, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - University Of Connecticut Health Center, Farmington, Connecticut
  - University Of Miami Center For Liver Diseases, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Rush University Med Ctr, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Medical Procare, Pllc, Flushing, New York
  - Office Of Sing Chan Md, Flushing, New York
  - Beth Israel Medical Center, New York, New York
  - Va New York Harbor Healthcare System, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Phgi Associates, Ltd, Philadelphia, Pennsylvania
  - Thomas Jefferson Medical College, Philadelphia, Pennsylvania
  - Upmc Center For Liver Diseases, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
- Argentina (7):
  - Local Institution, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution, El Palomar, Buenos Aires
  - Local Institution, San Salvador de Jujuy, Jujuy Province
  - Local Institution, Villa Nueva, Mendoza Province
  - Local Institution, Salta, Salta Province
  - Local Institution, Buenos Aires
  - Local Institution, Neuquén
- Brazil (24):
  - Local Institution, Rio Branco, Acre
  - Local Institution, Manaus, Amazonas
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Goiânia, Goiás
  - Local Institution, Cuiabá, Mato Grosso
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Ipatinga, Minas Gerais
  - Local Institution, Juiz de Fora, Minas Gerais
  - Local Institution, Curitiba, Paraná
  - Local Institution, Belém, Pará
  - Local Institution, Recife, Pernambuco
  - Local Institution, Rio de Janeiro / Rj, Rio de Janeiro
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Porto Alegres/rs, Rio Grande do Sul
  - Local Institution, São José, Santa Catarina
  - Local Institution, Campinas, São Paulo
  - Local Institution, Marília, São Paulo
  - Local Institution, Santo Andre - Sp, São Paulo
  - Local Institution, São José do Rio Preto, São Paulo
  - Local Institution, São Paulo, São Paulo
  - Local Institution, Sorocaba, São Paulo
  - Local Institution, Ribeirão Preto
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Canada (5):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- China (27):
  - Local Institution, Hefei, Anhui
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Chongqing, Chongqing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Shenzhen, Guangdong
  - Local Institution, Guiyang, Guizhou
  - Local Institution, Haikou, Hainan
  - Local Institution, Zhengzhou, Henan
  - Local Institution, Wuhan, Hubei
  - Local Institution, Changsha, Hunan
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Suzhou, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Dalian, Liaoning
  - Local Institution, Shenyang, Liaoning
  - Local Institution, Taiyuan, Shan1xi
  - Local Institution, Xi'an, Shan3xi
  - Local Institution, Jinan, Shandong
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Tianjin, Tianjin Municipality
  - Local Institution, Kunming, Yunnan
  - Local Institution, Hangzhou, Zhejiang
  - Local Institution, Linhai, Zhejiang
  - Local Institution, Ningbo, Zhejiang
  - Local Institution, Guangzhou
  - Local Institution, Shanghai
- Colombia (2):
  - Local Institution, Bogota, Cundinamarca
  - Local Institution, Bogotá
- Czechia (5):
  - Local Institution, Brno
  - Local Institution, Hradec Králové
  - Local Institution, Ostrava
  - Local Institution, Prague
  - Local Institution, Ústí nad Labem
- France (7):
  - Local Institution, Créteil
  - Local Institution, Grenoble
  - Local Institution, Lille
  - Local Institution, Limoges
  - Local Institution, Lyon
  - Local Institution, Paris
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (7):
  - Local Institution, Berlin
  - Local Institution, Bonn
  - Local Institution, Düsseldorf
  - Local Institution, Hamburg
  - Local Institution, Leipzig
  - Local Institution, Tübingen
  - Local Institution, Würzburg
- Greece (3):
  - Local Institution, Athens, Kolonaki
  - Local Institution, Alexandroupoli
  - Local Institution, Athens
- India (24):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Visakhapatnam, Andhra Pradesh
  - Local Institution, Secunderabad, Andhra Pradsh
  - Local Institution, Ahemedabad, Gujarat
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Gurgaon, Haryana
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Mangalore, Karnataka
  - Local Institution, Kochi, Kerala
  - Local Institution, Bhopal, Madhya Pradesh
  - Local Institution, Nagpur, Maharashtra
  - Local Institution, Nashik, Maharashtra
  - Local Institution, Ludhiana, Punjab
  - Local Institution, Jaipur, Rajasthan
  - Local Institution, Chennai, Tamil Nadu
  - Local Institution, Madurai, Tamil Nadu
  - Local Institution, Lucknow, Uttar Pradesh
  - Local Institution, Coimbatore
  - Local Institution, Hyderabad
  - Local Institution, Indore
  - Local Institution, Kolkata
  - Local Institution, Ludhiana
  - Local Institution, Mumbai
  - Local Institution, New Delhi
- Italy (3):
  - Local Institution, Bologna
  - Local Institution, Napoli
  - Local Institution, Rome
- Mexico (10):
  - Local Institution, Saltillo, Coahuila
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Cuernavaca, Morelos
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Monterrey, N.l., Nuevo León
  - Local Institution, Culiacan, Sin., Sinaloa
  - Local Institution, Boca del Rio, Veracruz
  - Local Institution, Distrito Federal
  - Local Institution, Durango
- Philippines (6):
  - Local Institution, Cebu City
  - Local Institution, Davao City
  - Local Institution, Ermita Manila
  - Local Institution, Manila
  - Local Institution, Metro Manila
  - Local Institution, Quezon City
- Poland (6):
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Poznan
  - Local Institution, Racibórz
  - Local Institution, Szczecin
  - Local Institution, Zawiercie
- Portugal (4):
  - Local Institution, Braga
  - Local Institution, Coimbra
  - Local Institution, Lisbon
  - Local Institution, Porto
- Romania (4):
  - Local Institution, Bucharest
  - Local Institution, Constanța
  - Local Institution, Iași
  - Local Institution, Timișoara
- Russia (12):
  - Local Institution, Kazan', Tatarstan Republic
  - Local Institution, Arkhangelsk
  - Local Institution, Irkutsk
  - Local Institution, Kirov
  - Local Institution, Krasnoyarsk
  - Local Institution, Lipetsk
  - Local Institution, Moscow
  - Local Institution, Nizhniy Novgord
  - Local Institution, Nizhny Novgorod
  - Local Institution, Ryazan
  - Local Institution, Samara
  - Local Institution, Yakutsk
- Local Institution, Singapore, Singapore
- South Korea (22):
  - Local Institution, Ansan-si, Gyeonggi-do
  - Local Institution, Uijeongbu-si, Gyeonggi-do
  - Local Institution, Bucheon-si
  - Local Institution, Busan
  - Local Institution, Chuncheon
  - Local Institution, Chungju
  - Local Institution, Daegu
  - Local Institution, Daejeon
  - Local Institution, Gangneung-si
  - Local Institution, Goyang
  - Local Institution, Gwangju
  - Local Institution, Gyeonggi-do
  - Local Institution, Gyeongju
  - Local Institution, Incheon
  - Local Institution, Jinju
  - Local Institution, Koyang City
  - Local Institution, Seoul
  - Local Institution, Sungnam-si
  - Local Institution, Sungnam
  - Local Institution, Suwon
  - Local Institution, Ulsan
  - Local Institution, Wŏnju
- Spain (6):
  - Local Institution, Granada
  - Local Institution, Madrid
  - Local Institution, Oviedo
  - Local Institution, San Sebastian Guipuzcuoa
  - Local Institution, Seville
  - Local Institution, Valencia
- Taiwan (5):
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Tainan
  - Local Institution, Taipei
  - Local Institution, Young Kang City
- Thailand (4):
  - Local Institution, Hat Yai, Changwat Songkhla
  - Local Institution, Bangkok
  - Local Institution, Khon Kaen
  - Local Institution, Pathum Thani
- Turkey (Türkiye) (6):
  - Local Institution, Adana
  - Local Institution, Ankara
  - Local Institution, Eskişehir
  - Local Institution, Izmir
  - Local Institution, Kayseri
  - Local Institution, Trabzon

REFERENCES:
- [Derived] Lim JK, Chang AY, Zaman A, Martin P, Fernandez-Rodriguez CM, Korkmaz M, Rossi S, Ford JM, Noonan T, Cooney E, Navarro V, Colombato L. Clinical Outcome Event Adjudication in a 10-Year Prospective Study of Nucleos(t)ide Analogue Therapy for Chronic Hepatitis B. J Clin Transl Hepatol. 2020 Dec 28;8(4):377-384. doi: 10.14218/JCTH.2020.00039. Epub 2020 Oct 10. PMID 33447520
- [Derived] Hou JL, Zhao W, Lee C, Hann HW, Peng CY, Tanwandee T, Morozov V, Klinker H, Sollano JD, Streinu-Cercel A, Cheinquer H, Xie Q, Wang YM, Wei L, Jia JD, Gong G, Han KH, Cao W, Cheng M, Tang X, Tan D, Ren H, Duan Z, Tang H, Gao Z, Chen S, Lin S, Sheng J, Chen C, Shang J, Han T, Ji Y, Niu J, Sun J, Chen Y, Cooney EL, Lim SG. Outcomes of Long-term Treatment of Chronic HBV Infection With Entecavir or Other Agents From a Randomized Trial in 24 Countries. Clin Gastroenterol Hepatol. 2020 Feb;18(2):457-467.e21. doi: 10.1016/j.cgh.2019.07.010. Epub 2019 Jul 12. PMID 31306800
- [Derived] Hou JL, Jia JD, Wei L, Zhao W, Wang YM, Cheng M, Tang X, Tan DM, Ren H, Tang H, Cohen D, Llamoso C. Efficacy and safety of entecavir treatment in a heterogeneous CHB population from a 'real-world' clinical practice setting in China. J Viral Hepat. 2013 Nov;20(11):811-20. doi: 10.1111/jvh.12115. PMID 23876210
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 12,522 participants were enrolled;12,485 participants were randomized; and12,378 participants received treatment. 100 participants were never treated with the study medication; 3 participants were at participant's request; 2 participants were not reported; 1 participant was administrative reason by sponsor; and 1 was other.
Groups:
- Entecavir (ETV): Tablets / Oral Solution, Oral, ETV = 0.5 mg - 1 mg, once daily.
- Other Anti-HBV Medication (Non-ETV): Standard of care HBV Nucleoside/Nucleotide Monotherapy, specific agent selected at the discretion of the investigator
Period: Initial Treatment
Arm/Group | Entecavir (ETV) | Other Anti-HBV Medication (Non-ETV)
Started | 6216 | 6162
Completed | 4388 (Completed=Reason of 'successful treatment', 'other: successful treatment' or 'other: end of study') | 3576 (Completed=discontinued initial treatment reason of "successful treatment" or "end of study")
Not Completed | 1828 | 2586
Not completed — Administrative Reason by Sponsor | 241 | 158
Not completed — Adverse Event | 22 | 87
Not completed — Death | 215 | 216
Not completed — Non-HCC HBV Disease Progression | 11 | 17
Not completed — HCC | 12 | 20
Not completed — Lost to Follow-up | 526 | 624
Not completed — Malignancy (Non-HCC) | 7 | 3
Not completed — Never Treated with Study Medication | 1 | 7
Not completed — Non-Study related Comorbidities | 3 | 4
Not completed — Not Defined | 125 | 172
Not completed — Partial or inadequate Treatment | 112 | 472
Not completed — Pregnancy | 26 | 16
Not completed — Study Drug Toxicity | 5 | 92
Not completed — Participant Request | 501 | 673
Not completed — No Off-Treatment Status Data | 11 | 13
Not completed — Not Reported | 10 | 12
Period: End of Study
Arm/Group | Entecavir (ETV) | Other Anti-HBV Medication (Non-ETV)
Started | 6216 | 6162
Completed | 4482 (Completed=Reason of 'other: end of study') | 3993 (Completed=Reason of 'other: end of study')
Not Completed | 1734 | 2169
Not completed — Administrative Reason By Sponsor | 299 | 253
Not completed — Death | 239 | 262
Not completed — HBV Disease Progression (Non-HCC) | 3 | 9
Not completed — HCC | 8 | 7
Not completed — Lost to Follow-up | 587 | 715
Not completed — Malignancy (Non-HCC) | 1 | 1
Not completed — Non-Study Related Comorbidities | 3 | 4
Not completed — Not Defined | 135 | 214
Not completed — Participant Withdrew Consent | 437 | 673
Not completed — No Off-Treatment Status Data | 22 | 30
Not completed — Not Reported | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Randomized Treated Subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Entecavir (ETV) | Other Anti-HBV Medication (Non-ETV) | Total
Number analyzed (Participants) | 6216 | 6162 | 12378
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (12.11) | 39.6 (12.14) | 39.7 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1503 | 1490 | 2993
  Male | 4713 | 4672 | 9385
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 153 | 154 | 307
  Unknown or Not Reported | 6060 | 6008 | 12068
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5221 | 5201 | 10422
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 59 | 68 | 127
  White | 819 | 780 | 1599
  Other | 113 | 111 | 224
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adjudicated Overall Malignant Neoplasms
Description: The number of participants with Overall Malignant Neoplasm, as adjudicated by Events Adjudication Committee (EAC)
Time Frame: 10 years
Population: All randomized, treated participants
Measure: Number; unit: Participants
Arm/Group | Entecavir (ETV) | Other Anti-HBV Medication (Non-ETV)
Number analyzed (Participants) | 6216 | 6162
Participants | 331 [0.800 to 1.084] | 337 [0.800 to 1.084]
Statistical Analysis 1: Comparison: Entecavir (ETV) vs Other Anti-HBV Medication (Non-ETV); Test type: Superiority or Other; p = 0.3553, Cox proportional hazards model; Hazard Ratio (HR) = 0.93, 95.03% CI 2-sided [0.800 to 1.084] — Hazard Ratio of ETV : Non-ETV Analyses are stratified by geographic region and prior HBV nucleoside/tide experience

2. Primary Outcome: Number of Deaths
Description: The number of deaths, as adjudicated by Events Adjudication Committee (EAC)
Time Frame: 10 years
Population: All randomized, treated participants
Measure: Number; unit: Participants
Arm/Group | Entecavir (ETV) | Other Anti-HBV Medication (Non-ETV)
Number analyzed (Participants) | 6216 | 6162
Participants | 238 [0.800 to 1.084] | 264 [0.800 to 1.084]
Statistical Analysis 1: Comparison: Entecavir (ETV) vs Other Anti-HBV Medication (Non-ETV); Test type: Superiority or Other; p = 0.0676, Cox proportional hazards model; Hazard Ratio (HR) = 0.85, 95.03% CI 2-sided [0.713 to 1.012] — Hazard Ratio of ETV : Non-ETV Analyses are stratified by geographic region and prior HBV nucleoside/tide experience

3. Primary Outcome: Number of Participants With Liver-related HBV Disease Progression
Description: The number of participants with Liver-related HBV disease progression, as adjudicated by Events Adjudication Committee (EAC)
Time Frame: 10 years
Population: All randomized, treated participants
Measure: Number; unit: Participants
Arm/Group | Entecavir (ETV) | Other Anti-HBV Medication (Non-ETV)
Number analyzed (Participants) | 6216 | 6162
Participants | 350 [0.800 to 1.084] | 375 [0.800 to 1.084]
Statistical Analysis 1: Comparison: Entecavir (ETV) vs Other Anti-HBV Medication (Non-ETV); Test type: Superiority or Other; p = 0.1182, Cox proportional hazards model; Hazard Ratio (HR) = 0.89, 95.03% CI 2-sided [0.769 to 1.030] — Hazard Ratio of ETV : Non-ETV Analyses are stratified by geographic region and prior HBV nucleoside/tide experience

4. Secondary Outcome: Number of Participants With Non-HCC Malignant Neoplasm
Description: The number of participants with non-HCC malignant neoplasm, as adjudicated by Events Adjudication Committee (EAC)
Time Frame: 10 years
Population: All randomized, treated participants
Measure: Number; unit: Participants
Arm/Group | Entecavir (ETV) | Other Anti-HBV Medication (Non-ETV)
Number analyzed (Participants) | 6216 | 6162
Participants | 95 [0.800 to 1.084] | 81 [0.800 to 1.084]
Statistical Analysis 1: Comparison: Entecavir (ETV) vs Other Anti-HBV Medication (Non-ETV); Test type: Superiority or Other; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.817 to 1.478] — Hazard Ratio of ETV : Non-ETV Analyses are stratified by geographic region and prior HBV nucleoside/tide experience

5. Secondary Outcome: Number of Participants With HCC Malignant Neoplasm
Description: The number of participants with HCC malignant neoplasm, as adjudicated by Events Adjudication Committee (EAC)
Time Frame: 10 years
Population: All randomized, treated participants
Measure: Number; unit: Participants
Arm/Group | Entecavir (ETV) | Other Anti-HBV Medication (Non-ETV)
Number analyzed (Participants) | 6216 | 6162
Participants | 240 [0.800 to 1.084] | 263 [0.800 to 1.084]
Statistical Analysis 1: Comparison: Entecavir (ETV) vs Other Anti-HBV Medication (Non-ETV); Test type: Superiority or Other; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.727 to 1.032] — Hazard Ratio of ETV : Non-ETV Analyses are stratified by geographic region and prior HBV nucleoside/tide experience

6. Secondary Outcome: Number of Participants With Liver-related Death
Description: The number of participants with Liver-related death, as adjudicated by Events Adjudication Committee (EAC)
Time Frame: 10 years
Population: All randomized, treated participants
Measure: Number; unit: Participants
Arm/Group | Entecavir (ETV) | Other Anti-HBV Medication (Non-ETV)
Number analyzed (Participants) | 6216 | 6162
Participants | 46 [0.800 to 1.084] | 48 [0.800 to 1.084]
Statistical Analysis 1: Comparison: Entecavir (ETV) vs Other Anti-HBV Medication (Non-ETV); Test type: Superiority or Other; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.608 to 1.365] — Hazard Ratio of ETV : Non-ETV Analyses are stratified by geographic region and prior HBV nucleoside/tide experience

ADVERSE EVENTS:
Time Frame: 10 years
Description: Mandatory reporting of non-serious AEs was not required. Reporting of serious adverse events (SAEs) which are considered unrelated (i.e. not likely or not related) to study drug was also not required.
Arm/Group | Entecavir (ETV) | Other Anti-HBV Medication (Non-ETV)
Serious Adverse Events (participants affected / at risk) | 56/6216 | 50/6162
Other Adverse Events (participants affected / at risk) | 0/6216 | 0/6162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entecavir (ETV) (N=6216) | Other Anti-HBV Medication (Non-ETV) (N=6162)
Ascites (Gastrointestinal disorders) | 3 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 0
Varices oesophageal (Gastrointestinal disorders) | 2 | 0
Chest discomfort (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Electrocution (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pelvic mass (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Chronic hepatitis (Hepatobiliary disorders) | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 2 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 4 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 0
Chronic hepatitis b (Infections and infestations) | 1 | 0
Hepatitis b (Infections and infestations) | 0 | 1
Hepatitis b reactivation (Infections and infestations) | 1 | 0
Tuberculous pleurisy (Infections and infestations) | 1 | 0
Atypical femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 3
Blood creatinine increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 4
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 15
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 2
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 0
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Coma hepatic (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Mononeuropathy (Nervous system disorders) | 0 | 1
Mononeuropathy multiplex (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 0 | 3
Nephropathy toxic (Renal and urinary disorders) | 0 | 2
Renal impairment (Renal and urinary disorders) | 1 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.